CLINICAL TRIAL: NCT07145177
Title: A Phase 1b Study of 177Lu-PSMA-617 Combined With Liver Directed Therapy in Metastatic Castration Resistant Prostate Cancer
Brief Title: 177Lu-PSMA-617 With Liver Directed Therapy in Metastatic Castration Resistant Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25929; NCI-2025-05994 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Prostate Cancer; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; Lutetium-177; Magnetic Resonance Spectroscopy; Biopsy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (177Lu-PSMA-617) (Experimental): Participants with diffusely PSMA-avid disease will receive standard doses of both 177Lu-PSMA-617 (7.4 Gigabequerel (GBq) every 6 weeks for up to 6 cycles) and transarterial chemoembolization (TACE) and/or ablation. Participants with one or more PSMA-negative liver lesions and PSMA-avid disease at all other sites will be treated with a single session of liver-directed therapy (either TACE or ablation) prior to initiation of 177Lu-PSMA-617 treatment. After cycle 2 of 177Lu-PSMA-617, participants who have extrahepatic stable disease/response but hepatic stable disease or progression per RECIST v1.1 will undergo liver-directed therapy. If clinically indicated and extrahepatic disease remains stable after cycle 3 of 177Lu-PSMA-617, participants may undergo a second course of liver-directed therapy. Participants will continue on study until progressive disease, study completion, unacceptable toxicity, or death.
  Interventions: Drug: 177Lu-PSMA-617; Procedure: Ablation; Procedure: Trans-arterial chemoembolization (TACE); Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT); Procedure: Tumor Biopsy; Other: Questionnaire

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Given intravenously (IV)
  Other Names: Lutetium-177 (177Lu)-PSMA-617
Procedure: Ablation — Undergo ablation
  Other Names: surgical ablation
Procedure: Trans-arterial chemoembolization (TACE) — Undergo TACE
  Other Names: TACE
Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT) — Undergo imaging
  Other Names: PET/CT
Procedure: Tumor Biopsy — Undergo biopsy
  Other Names: Biopsy
Other: Questionnaire — Participant will complete questionnaire
  Other Names: Quality of life questionnaire

SUMMARY:
This is an open label, single arm, phase 1b study to determine the safety of combining sequential Prostate-Specific Membrane Antigen (PSMA)-targeted 177Lu-PSMA-617 radionuclide therapy with liver-directed therapy in metastatic castrate-resistant prostate cancer (mCRPC) patients with liver metastases amenable to liver-directed therapy who have progressed on at least one prior androgen pathway inhibitor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety profile of 177Lu-PSMA-617 in combination with liver-directed therapy.

II. To determine the investigator-assessed objective response rate per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria in patients with mCRPC treated with 177LuPSMA-617 and liver-directed therapy.

SECONDARY OBJECTIVES:

I. To determine the median radiographic progression-free survival per PCWG3 criteria in patients with mCRPC treated with 177Lu-PSMA-617 and liver-directed therapy.

II. To determine the median overall survival in patients with mCRPC treated with 177Lu-PSMA-617 and liver-directed therapy.

III. To determine the median investigator-assessed duration of objective response per RECIST 1.1 criteria in patients with mCRPC treated with 177Lu-PSMA-617 and liver-directed therapy.

IV. To determine the investigator-assessed hepatic disease response rate (HDRR) per RECIST 1.1 in patients with mCRPC treated with 177Lu-PSMA-617 and liver-directed therapy.

V. To determine the investigator-assessed hepatic disease control rate (HDCR) at 6 months per RECIST 1.1 in patients with mCRPC treated with 177Lu-PSMA-617 and liver-directed therapy.

VI. To determine the PSA response rate by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria for participants with 50% decline (PSA50) and participants with a 90% decline (PSA90) at any time point on study, as well as individually following each dose of 177Lu-PSMA-617 or liver-directed therapy.

OUTLINE:

Participants will receive treatment with 177Lu-PSMA-617 for up to six total cycles every 6 weeks. Participants with one or more PSMA-negative liver lesions with a single session of liver-directed therapy prior to initiation of study drug. Participants will be follow-up every 3 months up to 5 years after the last study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate cancer.
2. Progressive disease by PCWG3 criteria at study entry.
3. Male participants who are at least 18 years of age on the day of signing informed consent.
4. Castrate level of serum testosterone at study entry (< 50 ng/dL). Note: Participants without prior bilateral orchiectomy are required to remain on Luteinizing hormone-releasing hormone (LHRH) analogue treatment for duration of study treatment.
5. Prior progression on at least one second generation androgen signaling inhibitor including abiraterone, apalutamide, darolutamide, and/or enzalutamide.
6. Adverse events related to prior anti-cancer treatment (excluding LHRH analogs) must have recovered to Grade ≤ 1 (except for any grade alopecia and grade ≤ 2 neuropathy).
7. Prior external beam radiotherapy is allowed if the last radiotherapy treatment was greater than 2 weeks from start of study treatment on Cycle 1 Day 1 (C1D1). Note: Participants must have recovered from all radiation-related toxicities. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
8. At least one PSMA-avid extrahepatic lesion on screening PSMA Positron Emission Tomography (PET). A positive lesion is defined as uptake above background liver. Hepatic lesions may be PSMA PETnegative or positive.
9. Availability of archival mCRPC tissue, or presence of a metastatic lesion that is amenable to fresh biopsy and willingness to undergo biopsy during screening if no archival mCRPC tissue available.
10. The presence of one or more liver metastases amenable to liver-directed therapy in the judgment of the treating interventional radiologist. Liver metastases may be detected by CT or magnetic resonance imaging (MRI), and biopsy confirmation is not required.
11. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 or Karnofsky ≥ 50%.
12. Demonstrates adequate organ function as defined below:

    1. Absolute neutrophil count ≥ 1,500/ microliter (mcL).
    2. Platelets ≥ 100,000/mcL.
    3. Hemoglobin > 9.0 g/dL.
    4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN). In participants with known or suspected Gilbert's disease, direct bilirubin ≤ ULN.
    5. aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) ≤ 5 x institutional upper limit of normal.
    6. alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) ≤ 5 x institutional upper limit of normal.
    7. Prothrombin time ≤ 1.5 x institutional upper limit of normal (unless on medical therapy known to prolong prothrombin time).
    8. Albumin ≥ 2.8 g/dL
    9. Creatinine clearance Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2, calculated using the Cockcroft-Gault equation or 24 hour urine collection.
13. Participants with previously treated brain metastases are eligible provided the following criteria are all met:

    1. Last treatment was > 28 days prior to C1D1
    2. No evidence of new/progressive brain metastases is observed on MRI obtained during the Screening window
14. Participants must use appropriate methods of contraception during study treatment and for at least 6 months after last study treatment. Note: Participants who are sexually active should consider their female partner to be of childbearing potential if she has experienced menarche and is not postmenopausal (defined as amenorrhea > 24 consecutive months) or has not undergone successful surgical sterilization. Even women who use contraceptive hormones (oral, implanted, or injected), an intrauterine device, or barrier methods (diaphragms, condoms, spermicide) should be considered to be of childbearing potential. Participants who have undergone vasectomy themselves should also be considered to be of childbearing potential. Acceptable methods of contraception include continuous total abstinence, or double barrier method of birth control (e.g., condoms used with spermicide, or condoms used with oral contraceptives). Periodic abstinence and withdrawal are not acceptable methods of contraception.
15. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. De novo small cell neuroendocrine prostate cancer.
2. One or more extrahepatic soft tissue lesions (lymph nodes > 1.5 cm in short axis, visceral/soft tissue lesions > 1 cm) on screening CT that is negative on PSMA PET. Non- PSMA avid liver lesions are allowed.
3. Recipient of other systemic anti-cancer therapies administered within 14 days, or 5 half lives, whichever is shorter, prior to initiation of study treatment. Note: LHRH analogues are the exception and are permitted
4. Recipient of prior PSMA-directed radioligand treatment.
5. Recipient of > 2 lines of prior taxane-based chemotherapy administered in the castration-resistant setting. Prior taxane in the castration sensitive setting does not count towards this limit. If platinum chemotherapy is added to taxane this does not count as a separate line of treatment.
6. Previous bilio-enteric anastomosis, ampulla of Vater sphincterotomy, biliary stent, or biliary drain passing through the ampulla of Vater.
7. Currently participating in a study of an investigational therapeutic agent or has used an investigational device within 4 weeks prior to the first dose of study treatment on C1D1. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
8. Clinically significant cardiovascular disease including, but not limited to:

   1. Uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure.
   2. Uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months before study entry.
   3. Clinically significant arrhythmias not controlled by medication. Note: Chronic rate-controlled or paroxysmal atrial fibrillation/flutter is not an exclusion to study participation.
9. Major surgery within 28 days of study treatment. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment on C1D1. Minor procedures (e.g., biopsy, cataract surgery, stent placement, endoscopy) are not considered major surgery.
10. Has a secondary malignancy requiring active treatment at study entry (except for carcinoma-in-situ, non-muscle invasive bladder cancer, and non-melanoma skin cancer).
11. Has an active infection requiring intravenous antibiotics within 7 days prior to C1D1.
12. Has a known history of Hepatitis B infection (Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection (HCV RNA [qualitative] detected, with the following exceptions:

    1. Participants who are HbsAg positive are eligible if they have received hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to study entry.
    2. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening. Participants must have completed curative anti-viral therapy at least 4 weeks prior to study entry.
13. Not a candidate for liver-directed therapy on the basis of any of the following:

    1. History of bleeding diathesis and currently on anti-coagulation therapy that cannot be safely discontinued for liver directed therapy.
    2. Clinically significant ascites including requiring more than one paracentesis in the 28 days prior to C1D1.
14. Unable or unwilling to follow radiation safety precautions following each dose of radioligand therapy or liver directed therapy.
15. Any condition that, in the opinion of the Principal Investigator, would impair the participant's ability to comply with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment emergent adverse events. | up to 12 months
  Treatment emergent adverse events will be classified according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Adverse events and clinically significant laboratory abnormalities (meeting Grade 3, 4, or 5 criteria according to CTCAE) will be summarized by maximum intensity and relationship to Lu-PSMA-617 and liver-directed therapy (if applicable). Descriptive statistics will be utilized to display the data on toxicity seen. Descriptive summaries of discrete data will present the number of study participants and the incidence as a frequency and a percentage.
Objective response Rate (ORR) | up to 12 months
  ORR is defined as the proportion of treated participants who obtained an radiographic objective response [confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Proportion and 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Median radiographic Progression-free survival (rPFS) | up to 12 months
  rPFS is defined as the time that elapses between the initiation of trial therapy Cycle 1 Day 1(C1D1) and the date of radiographic disease progression per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria for all evaluable patients. If disease progression or death from any cause is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the rPFS will be censored as the last available disease assessment. Patients who discontinue treatment for clinical progression or deterioration will be included in the analysis. Calculated based on Kaplan-Meier estimates of rPFS.
Median Overall Survival (OS) | up to 5 years
  OS is defined as the overall survival time as the time that elapses between the initiation of trial therapy C1D1 and the date of death from any cause for all evaluable patients. Calculated based on Kaplan-Meier estimates of OS.
Median duration of objective response (mDOR) | up to 12 months
  mDOR is defined as the time that elapses between the day of first documented response to trial therapy (confirmed CR or confirmed PR, whichever is first recorded) and subsequent disease progression (per RECIST v1.1 criteria). Results will be calculated based on Kaplan-Meier product limit method.
Hepatic disease response rate (HDRR) | up to 12 months
  HDRR is defined as the proportion of treated patients who experience an objective hepatic response [confirmed complete response (CR) or confirmed partial response (PR) per RECIST v1.1criteria.
Hepatic disease control rate (HDCR) | 6 months
  HDCR is defined as the proportion of treated patients who experience 6 months of hepatic disease control from the day of first documented hepatic response to trial therapy (confirmed CR or confirmed PR, whichever is first recorded) per RECIST v1.1criteria, until hepatic disease progression, change in anti-cancer therapy, or study completion.
Proportion of Participants With a >=50% Decline in Prostate Specific Antigen (PSA) | up to 15 months
  The proportion of participants who achieve greater than 50% decline in baseline PSA (baseline drawn on C1D1), at any point during treatment. Proportion and 95% confidence interval will be reported.
Proportion of Participants With a >=90% Decline in PSA | up to 15 months
  The proportion of participants who achieve greater than 90% decline in baseline PSA (baseline drawn on C1D1), at any point during treatment. Proportion and 95% confidence interval will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No